CLINICAL TRIAL: NCT01761084
Title: Build Better Bones With Exercise: A Pilot Randomized Controlled Trial of Exercise in Women With Osteoporotic Vertebral Fracture
Brief Title: Build Better Bones With Exercise
Acronym: B3E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Western Ontario, Canada (Other); University Health Network, Toronto (Other); McMaster University (Other); University of Melbourne (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18539
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2017-03

CONDITIONS: Osteoporotic Fractures; Spinal Fractures
Keywords: Osteoporosis; Spine fracture; Vertebral fracture; Exercise Interventions; Exercise
MeSH Terms: conditions — Osteoporotic Fractures; Spinal Fractures; Osteoporosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise and behaviour change strategies (Experimental): The exercise program will include strength training, balance training and cardiovascular exercise that is individually tailored to the participants' abilities. The physical therapist will also implement strategies to assist with behaviour change, such as documenting progress in a log, participating in action planning and coping planning, and using techniques in the spirit of motivational interviewing.
  Interventions: Behavioral: Exercise and behaviour change strategies
- General health or social discussion (No Intervention): Participants in the control group will receive equal attention, but will not be prescribed exercise, or participate in counselling about exercise. The physical therapist will discuss topics related to general health.

INTERVENTIONS:
Behavioral: Exercise and behaviour change strategies — 1. cardiovascular exercise (e.g., marching, walking) for ≥10 minutes per day
  2. postural retraining and balance exercises ≥3 days a week (will be encouraged to do these daily)
  3. perform muscle strengthening and balance training exercises ≥ 3 days a week
  4. the exercise intervention was developed using the Bone Fit program as a framework (http://www.bonefit.ca/). The physical therapist will tailor exercises and work with participant to integrate them into their day.
  Arms: Exercise and behaviour change strategies

SUMMARY:
The long-term goal of our research team is to conduct a large multicentre study to evaluate whether tailored home exercise can prevent fractures in high-risk individuals. The proposed project will address the feasibility of such a trial, but will also evaluate the effect of exercise on quality of life, posture and many other outcomes important to individuals with vertebral fractures. Physiotherapists will conduct 6 home visits with participants to deliver the intervention (or social visit for controls) using a similar model to previous work by our team and others. The purpose of this pilot study is determining the feasibility of recruitment, retention and adherence of an international multicentre randomized controlled study evaluating the efficacy of thrice-weekly home exercise for one year among women with vertebral fracture. As secondary objectives, the investigators will examine the effects of exercise on function, balance, quality of life, pain, falls and fractures. The primary hypothesis is that the investigators will successfully recruit and retain the target sample, and achieve an adherence rate of 60%.

DETAILED DESCRIPTION:
There is limited data available from which to develop guidelines for safe and effective exercise prescription among individuals with hip or vertebral fractures. The long-term goal of our research team is to conduct a large multi-centre randomized controlled trial (RCT) to investigate whether participating in a thrice-weekly home exercise program for one year can reduce incident fragility fractures among women aged 65 years or older with a history of vertebral fracture compared to no intervention. The current study is a pilot study with the principal objective of determining the feasibility of recruitment, retention and adherence of an international multicentre RCT evaluating the efficacy of thrice-weekly home exercise for one year among women with vertebral fracture. The intervention was developed by experts in exercise prescription based on a rigorous literature review and Cochrane meta-analysis we have conducted. Physiotherapists will conduct 6 home visits with participants to deliver the intervention (or social visit for controls) using a similar model to previous work by our team and others. Secondary outcomes of the pilot study are those hypothesized to be among the causal pathway linking exercise to fracture risk, including lower extremity strength, posture, balance, as well as falls and fractures. Additional secondary outcomes include quality of life, pain, exercise self-efficacy, the cost of the intervention, and the risk of adverse events associated with exercise. The recruitment and retention process will be summarized using a CONSORT flow diagram, and the reporting of results will be in accordance with the CONSORT criteria. Analyses of feasibility objectives will be descriptive or based on estimates with 95% confidence intervals, where feasibility will be assessed relative to criteria defined a priori. Differences in secondary outcomes will be evaluated in intention to treat analyses via independent student T-tests, Chi Square or logistic regression. The Bonferroni method will be used to adjust the level of significance for secondary outcomes so the overall level is alpha=0.05. Even if the larger trial proves not to be feasible, the current trial will be one of the largest exercise studies among a representative group of women with vertebral fracture to date, and will evaluate the feasibility and costs of a comprehensive home exercise program, and its effect on important secondary outcomes. Osteoporosis Canada has defined a need to develop patient resources on exercise and recently announced a shift in priority to individuals with existing fractures; the proposed pilot study is timely and will directly inform these knowledge translation initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Has a) a known or suspected vertebral fracture of non-traumatic etiology OR b) one of the following:

  * documented height loss of ≥2cm
  * historical height loss of ≥6cm
  * visible hyperkyphosis
* age greater than or equal to 65 years of age
* able to understand instructions in english
* able to give informed consent (no cognitive impairment)

Exclusion Criteria:

* Current or prior cancer
* On dialysis, known liver, kidney or malabsorption disease
* Progressive neurological disorder, unable to stand or walk for 10 metres, with/without gait aid or progressive disorder likely to prevent study completion, palliative care.
* Current participation in muscle strengthening or similar exercise program ≥ 3 times per week
* Uncontrolled hypertension or other contraindications to exercise

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 141 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lora Giangregorio, PhD, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

REFERENCES:
- [Derived] Gibbs JC, McArthur C, Wark JD, Thabane L, Scherer SC, Prasad S, Papaioannou A, Mittmann N, Laprade J, Kim S, Khan A, Kendler DL, Hill KD, Cheung AM, Bleakney R, Ashe MC, Adachi JD, Giangregorio LM. The Effects of Home Exercise in Older Women With Vertebral Fractures: A Pilot Randomized Controlled Trial. Phys Ther. 2020 Apr 17;100(4):662-676. doi: 10.1093/ptj/pzz188. PMID 31899499
- [Derived] Giangregorio LM, Thabane L, Adachi JD, Ashe MC, Bleakney RR, Braun EA, Cheung AM, Fraser LA, Gibbs JC, Hill KD, Hodsman AB, Kendler DL, Mittmann N, Prasad S, Scherer SC, Wark JD, Papaioannou A. Build better bones with exercise: protocol for a feasibility study of a multicenter randomized controlled trial of 12 months of home exercise in women with a vertebral fracture. Phys Ther. 2014 Sep;94(9):1337-52. doi: 10.2522/ptj.20130625. Epub 2014 May 1. PMID 24786946
- See also: Principal Investigator — https://uwaterloo.ca/kinesiology/people-profiles/lora-giangregorio

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise and Behaviour Change Strategies: The exercise program will include strength training, balance training and cardiovascular exercise that is individually tailored to the participants' abilities. The physical therapist will also implement strategies to assist with behaviour change, such as documenting progress in a log, participating in action planning and coping planning, and using techniques in the spirit of motivational interviewing.
  Exercise and behaviour change strategies: a)cardiovascular exercise (e.g., marching, walking) for ≥10 minutes per day b)postural retraining and balance exercises ≥3 days a week (will be encouraged to do these daily) c)perform muscle strengthening and balance training exercises ≥ 3 days a week d)the exercise intervention was developed using the Bone Fit program as a framework (http://www.bonefit.ca/). The physical therapist will tailor exercises and work with participant to integrate them into their day.
Period: Overall Study
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Started | 71 | 70
Completed | 66 | 64
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion | Total
Number analyzed (Participants) | 71 | 70 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (6.4) | 77 (7.28) | 76 (6.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 70 | 141
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment and Retention
Description: Number of participants recruited and retained. Criteria for success = 20 recruited per site and at least 75% retained.
Time Frame: Monthly records up to 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
Participants | 66 | 64

2. Primary Outcome: Adherence
Description: Number of exercise sessions completed relative to prescribed. We will use a diary for participants to self-report adherence.
Time Frame: Monthly records over 12 months
Population: Only the Exercise Group received the exercise program.
Measure: Mean (Full Range); unit: % of weeks meeting adherence threshold
Arm/Group | Exercise and Behaviour Change Strategies
Number analyzed (Participants) | 71
% of weeks meeting adherence threshold | 66 [17 to 86]

3. Secondary Outcome: Number of Fractures.
Description: Incident fracture will be a composite outcome of a vertebral fracture or fragility fracture (excluding fractures due to trauma or cancer). A fracture questionnaire will be used to ascertain the occurrence of fractures, the approximate timing and the cause with fracture occurrence, location and severity verified through health record data. Lateral thoracic and lumbar spine x-rays will be performed on participants at baseline (to confirm prevalent vertebral fractures) and follow-up (to identify new fractures). Vertebral fractures will be defined as radiographic presence of ≥25% reduction in anterior, middle or posterior height of a vertebra using the Genant visual semi-quantitative method.
Time Frame: Baseline, one year and at report of fracture (monitored monthly for reports).
Measure: Number; unit: Fractures
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
Fractures
  Baseline | 168 | 163
  12 Month Follow-up | 183 | 178
Statistical Analysis 1: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Test type: Superiority; Odds Ratio (OR) = 1.06, 95% CI 2-sided [.58 to 1.94]

4. Secondary Outcome: Number of Fallers
Description: Diary for participants to self-report falls.
Time Frame: Monthly up to one year.
Measure: Count of Participants; unit: Participants
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
Participants | 48 | 36
Statistical Analysis 1: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Test type: Superiority; Risk Ratio (RR) = 1.32, 95% CI 2-sided [.99 to 1.74]

5. Secondary Outcome: Occiput to Wall Distance
Time Frame: Baseline and one year.
Measure: Mean (Standard Deviation); unit: centimetres
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
centimetres
  Baseline | 5.3 (4.0) | 6.2 (4.7)
  Month 12 | 5.3 (4.4) | 6.1 (3.9)
Statistical Analysis 1: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Baseline; Test type: Superiority; p = 0.811, t-test, 2 sided; Intention-to-treat analysis; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.84 to 1.07] — Intention-to-treat analysis
Statistical Analysis 2: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Month 12; Test type: Superiority; p = 0.765, t-test, 2 sided; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.80 to 1.09] — Per-protocol analysis

6. Secondary Outcome: Scores on the Short Physical Performance Battery (SPPB)
Description: The SPPB consists of balance tests (side-by-side, semi-tandem, and tandem standing), gait speed during 4-meter walk test, and the average time taken to rise from a chair with arms folded across chest and sit back down (Five-Times-Sit-to-Stand test), sub-scores of which are added to determine a composite score (0-12), with higher scores indicative of better performance.
Time Frame: Baseline and one year.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
score on a scale
  Baseline | 9.6 (2.2) | 8.8 (2.3)
  12 months | 9.7 (2.5) | 9.0 (2.3)
Statistical Analysis 1: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Baseline; Test type: Superiority; p = 0.796, t-test, 2 sided; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.80 to 0.61] — Intention-to-treat analysis
Statistical Analysis 2: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Month 12; Test type: Superiority; p = 0.888, t-test, 2 sided; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.75 to 0.65] — Per-protocol analysis

7. Secondary Outcome: Scores on Balance Outcome Measure for Elder Rehabilitation (BOOMER).
Description: Balance Outcome Measure for Elder Rehabilitation (BOOMER) includes the step test, the Timed Up and Go, the Functional Reach test and the timed static stance feet together eyes closed test. The sub-scores of which are added to create a composite score (0-16), with higher scores indicating better performance.
Time Frame: Baseline and one year.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
score on a scale
  Baseline | 13.5 (2.2) | 13.2 (2.0)
  Month 12 | 13.6 (2.6) | 13.2 (2.3)
Statistical Analysis 1: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Baseline; Test type: Superiority; p = 0.719, t-test, 2 sided; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.54 to 0.78] — Intention-to-treat analysis
Statistical Analysis 2: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Month 12; Test type: Superiority; p = 0.745, t-test, 2 sided; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.56 to 0.79] — Per-protocol analysis

8. Secondary Outcome: Quality of Life (QoL) and Pain Scores Measured Through the EuroQOL Instrument (EQ5D5L) and the Osteoporosis Quality of Life Questionnaire (OQLQ) and a Visual Analog Scale (VAS).
Description: OQLQ scores range 1-7, with higher scores indicate greater quality of life. EQ5D5L VAS scores range 0-100, with higher scores indicating better overall health. VAS pain scores range 0-10, with lower scores indicating less pain.
Time Frame: Baseline, 6 months and one year.
Population: Withdrawals at 6 months - intervention group (n=4) and control group (n=5). Withdrawals at 12 months - intervention group (n=5) and control group (n=6).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
score on a scale
  EQ5D-VAS - Baseline | 74.1 (19.1) | 75.7 (20.0)
  EQ5D-VAS - Month 6: number analyzed (Participants) | 67 | 65
  EQ5D-VAS - Month 6 | 75.5 (17.6) | 75.7 (18.8)
  EQ5D-VAS - Month 12: number analyzed (Participants) | 66 | 64
  EQ5D-VAS - Month 12 | 74.6 (19.1) | 75.7 (15.4)
  OQLQ - Average - Baseline | 5.1 (1.3) | 5.2 (1.2)
  OQLQ - Average - Month 6: number analyzed (Participants) | 67 | 65
  OQLQ - Average - Month 6 | 5.4 (1.2) | 5.6 (1.2)
  OQLQ - Average - Month 12: number analyzed (Participants) | 66 | 64
  OQLQ - Average - Month 12 | 5.4 (1.4) | 5.4 (1.3)
  Pain VAS at Rest - Baseline | 2.7 (2.7) | 2.4 (2.1)
  Pain VAS at Rest - Month 6: number analyzed (Participants) | 67 | 65
  Pain VAS at Rest - Month 6 | 2.3 (2.4) | 2.1 (2.1)
  Pain VAS at Rest - Month 12: number analyzed (Participants) | 66 | 64
  Pain VAS at Rest - Month 12 | 1.9 (2.2) | 2.1 (2.2)
  Pain VAS Movement - Baseline | 3.8 (2.9) | 4.2 (2.6)
  Pain VAS Movement - Month 6: number analyzed (Participants) | 67 | 65
  Pain VAS Movement - Month 6 | 3.0 (2.4) | 3.5 (2.5)
  Pain VAS Movement - Month 12: number analyzed (Participants) | 66 | 64
  Pain VAS Movement - Month 12 | 3.6 (2.7) | 3.9 (2.5)
Statistical Analysis 1: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Comparison of change from baseline in EQ5D - VAS; Test type: Superiority; p = 0.854, t-test, 2 sided; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [-5.66 to 6.83] — Intention-to-treat analysis
Statistical Analysis 2: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Comparison of change from baseline in EQ5D-VAS; Test type: Superiority; p = 0.585, t-test, 2 sided; Mean Difference (Final Values) = 1.78, 95% CI 2-sided [-4.66 to 8.22] — Per-protocol analysis
Statistical Analysis 3: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Comparison of change from baseline in OQLQ Average Score; Test type: Superiority; p = 0.335, t-test, 2 sided; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.16 to 0.47] — Intention-to-treat analysis
Statistical Analysis 4: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Comparison of change from baseline in OQLQ Average Score; Test type: Superiority; p = 0.285, t-test, 2 sided; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.15 to 0.50] — Per-protocol analysis
Statistical Analysis 5: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Comparison of change from baseline in pain VAS at rest; Test type: Superiority; p = 0.225, t-test, 2 sided; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.36 to 0.32] — Intention-to-treat analysis
Statistical Analysis 6: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Comparison of change from baseline in pain VAS at rest; Test type: Superiority; p = 0.488, t-test, 2 sided; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-1.16 to 0.56] — Per-protocol analysis
Statistical Analysis 7: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Comparison of change from baseline in pain VAS during movement; Test type: Superiority; p = 0.808, t-test, 2 sided; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.68 to 0.88] — Intention-to-treat analysis
Statistical Analysis 8: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Comparison of change from baseline in pain VAS during movement; Test type: Superiority; p = 0.566, t-test, 2 sided; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.57 to 1.04] — Per-protocol analysis

9. Secondary Outcome: Scores on Exercise Self-efficacy Scales.
Description: To assess self-efficacy related to engaging in exercise, participants will be asked "Over the next 3 months, how confident are you that you can perform exercise on most days of the week?" and "Over the next 3 months, how confident are you that you can perform exercise on 3 days of the week?." To assess implementation intentions, participants are asked "Do you already have concrete plans regarding exercise?". Patients will rate their answers on a scale from 1-5. Higher scores indicate greater exercise self-efficacy.
Time Frame: Baseline, 6 months and one year.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
units on a scale
  Baseline | 4.4 (0.7) | 4.4 (0.6)
  Month 6: number analyzed (Participants) | 67 | 65
  Month 6 | 4.2 (0.7) | 4.0 (0.8)
  Month 12: number analyzed (Participants) | 66 | 64
  Month 12 | 4.0 (0.8) | 4.0 (0.7)

10. Secondary Outcome: Score on Short-form Falls Efficacy Scale International (FES-I).
Description: Questionnaire about how concerned the participant is about the possibility of falling during common daily activities. Scores range from 7 (no concern about falling) to 28 (severe concern about falling.
Time Frame: Baseline, 6 months and one year.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
score on a scale
  Baseline | 12.1 (4.8) | 12.9 (5.6)
  Month 6: number analyzed (Participants) | 67 | 65
  Month 6 | 11.4 (4.0) | 11.5 (4.7)
  Month 12: number analyzed (Participants) | 66 | 64
  Month 12 | 11.5 (4.7) | 12.3 (5.0)

11. Secondary Outcome: Productivity
Description: Questionnaire regarding much did the participant's spine fracture(s) or osteoporosis affect their productivity while working? The scale is 0-10, with higher numbers indicating more effect on their work.
Time Frame: Monthly up to one year.
Population: Only participants who reported working and/or volunteering were asked this question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
units on a scale
  Baseline: number analyzed (Participants) | 19 | 20
  Baseline | 1.89 (2.536) | 1.85 (1.927)
  Month 1: number analyzed (Participants) | 20 | 17
  Month 1 | 1.60 (2.257) | 1.76 (1.985)
  Month 2: number analyzed (Participants) | 19 | 17
  Month 2 | 1.32 (2.212) | 2.12 (1.965)
  Month 3: number analyzed (Participants) | 19 | 17
  Month 3 | 1.21 (2.149) | 2.94 (2.947)
  Month 4: number analyzed (Participants) | 18 | 18
  Month 4 | 1.00 (1.910) | 2.50 (2.307)
  Month 5: number analyzed (Participants) | 18 | 14
  Month 5 | 0.11 (.471) | 1.57 (1.910)
  Month 6: number analyzed (Participants) | 16 | 17
  Month 6 | 0.69 (1.778) | 1.88 (2.261)
  Month 7: number analyzed (Participants) | 15 | 14
  Month 7 | .80 (1.781) | 2.07 (2.556)
  Month 8: number analyzed (Participants) | 14 | 16
  Month 8 | 0.93 (2.056) | 2.00 (2.191)
  Month 9: number analyzed (Participants) | 14 | 17
  Month 9 | 1.07 (2.556) | 1.76 (2.333)
  Month 10: number analyzed (Participants) | 20 | 17
  Month 10 | 0.95 (2.089) | 1.24 (1.855)
  Month 11: number analyzed (Participants) | 16 | 18
  Month 11 | 0.88 (2.029) | 1.83 (2.503)
  Month 12: number analyzed (Participants) | 21 | 19
  Month 12 | 0.76 (2.022) | 2.16 (2.115)
Statistical Analysis 1: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Baseline; Test type: Superiority; p = .951, t-test, 2 sided; Mean Difference (Final Values) = 0.045, 95% CI 2-sided [-1.412 to 1.501]
Statistical Analysis 2: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Month 12; Test type: Superiority; p = 0.039, t-test, 2 sided; Mean Difference (Final Values) = -1.396, 95% CI 2-sided [-2.721 to -0.071]

12. Secondary Outcome: Physical Activity
Description: A modified version of the Short-Form International Physical Activity Questionnaire (IPAQ) will be completed. A subset of participants at the University of Waterloo (St. Mary's General Hospital) will wear an accelerometer for 7 days.
Time Frame: Baseline, 6 months, 12 months
Population: Withdrawals at 6 months - intervention group (n=4) and control group (n=5) Withdrawals at 12 months - intervention group (n=5) and control group (n=6)
Measure: Mean (Standard Deviation); unit: Minutes per week
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
Minutes per week
  Baseline Strength/Balance physical activity | 6.7 (17.0) | 6.4 (16.8)
  Baseline Moderate-Vigorous physical activity | 43.2 (138.5) | 48.8 (156.1)
  Baseline Walking | 168.8 (366.0) | 194.9 (278.3)
  Month 6 Strength/Balance physical activity: number analyzed (Participants) | 67 | 65
  Month 6 Strength/Balance physical activity | 80.8 (85.8) | 15.7 (36.4)
  Month 6 Moderate-Vigorous physical activity: number analyzed (Participants) | 67 | 65
  Month 6 Moderate-Vigorous physical activity | 76.1 (143.9) | 147.3 (346.0)
  Month 6 Walking: number analyzed (Participants) | 67 | 65
  Month 6 Walking | 165.4 (120.6) | 154.0 (161.6)
  Month 12 Strength/Balance physical activity: number analyzed (Participants) | 66 | 64
  Month 12 Strength/Balance physical activity | 68.4 (68.3) | 21.1 (44.9)
  Month 12 Moderate-Vigorous physical activity: number analyzed (Participants) | 66 | 64
  Month 12 Moderate-Vigorous physical activity | 93.9 (225.9) | 128.9 (352.3)
  Month 12 Walking: number analyzed (Participants) | 66 | 64
  Month 12 Walking | 161.2 (140.7) | 268.0 (342.3)
Statistical Analysis 1: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Only Month 6 and Month 12 strength and balance physical activity differences were significant; Test type: Superiority; p < 0.05, t-test, 2 sided — Month 6 strength and balance physical activity; Mean Difference (Final Values) = -65.9, 95% CI 2-sided [-91.8 to -40.0]
Statistical Analysis 2: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Only Month 6 and Month 12 strength and balance physical activity differences were significant; Test type: Superiority; p < 0.05, t-test, 2 sided — Month 12 strength and balance physical activity; Mean Difference (Final Values) = -49.3, 95% CI 2-sided [-69.8 to -28.8]

13. Secondary Outcome: Number of Serious Adverse Events.
Description: Defined as death or event that is life-threatening, requires hospitalization or results in disability.
Time Frame: Monthly up to one year.
Measure: Number; unit: events
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
events | 18 | 12

14. Secondary Outcome: Number of Individuals Screened and Eligible Per Collection Site.
Description: Number of participants randomized out of all participants screened
Time Frame: over the course of the study (2.29 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Screened
Number analyzed (Participants) | 2822
Participants | 141

15. Secondary Outcome: Number of Potentially Eligible Males
Time Frame: over recruitment period
Population: Total people screened for inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Screened
Number analyzed (Participants) | 2254
Participants | 308

16. Secondary Outcome: Number of Participants With Multiple Falls
Time Frame: Monthly up to 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
Participants | 31 | 22

17. Secondary Outcome: Total Number of Falls
Time Frame: Monthly up to 12 months.
Measure: Number; unit: Falls
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
Falls | 130 | 127
Statistical Analysis 1: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Negative Binomial Regression; Test type: Superiority; Incident Rate Ratio = .97, 95% CI 2-sided [.58 to 1.63]

18. Secondary Outcome: Value of Direct Medical Resources Per Participant.
Time Frame: Accrued costs over 12 months
Population: For each resource cost, only participants utilizing the resource are included.
Measure: Mean (Standard Deviation); unit: Dollars (Canadian)
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
Dollars (Canadian)
  Medications: number analyzed (Participants) | 71 | 67
  Medications | 2127 (3579) | 1823 (3063)
  Medical costs related to adverse events: number analyzed (Participants) | 35 | 23
  Medical costs related to adverse events | 1680 (3600) | 3130 (3180)
  Physician visits and tests/ procedures: number analyzed (Participants) | 65 | 62
  Physician visits and tests/ procedures | 829 (1033) | 848 (863)
  Allied health professional visits: number analyzed (Participants) | 5 | 4
  Allied health professional visits | 301 (331) | 95 (51)

19. Secondary Outcome: Value of Non-direct Medical Resources Per Participant.
Time Frame: Accrued costs over 12 months
Population: For each resource cost, only participants utilizing the resource are included.
Measure: Mean (Standard Deviation); unit: Dollars (Canadian)
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
Dollars (Canadian)
  Unpaid caregiver time: number analyzed (Participants) | 50 | 52
  Unpaid caregiver time | 5005 (9220) | 4631 (8091)
  Lost productivity: number analyzed (Participants) | 26 | 17
  Lost productivity | 998 (1642) | 917 (1322)
  Out of pocket costs: number analyzed (Participants) | 57 | 52
  Out of pocket costs | 1007 (1453) | 872 (1250)

20. Secondary Outcome: Participant Height
Time Frame: Baseline and one year
Population: Withdrawals at 12 months - intervention group (n=5) and control group (n=6). The remainder (5 intervention, 2 control) did not attend the follow-up visit.
Measure: Mean (Standard Deviation); unit: centimetres
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
centimetres
  Baseline | 156.5 (6.4) | 156.1 (7.2)
  Month 12: number analyzed (Participants) | 61 | 62
  Month 12 | 156.4 (6.6) | 155.9 (7.2)
Statistical Analysis 1: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Comparison of change from baseline in height; Test type: Superiority; p = 0.536, t-test, 2 sided; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.28 to 0.53] — Intention-to-treat analysis

21. Secondary Outcome: Activities of Daily Living
Description: 0-10 scale about ability to do activities of daily living. Higher scores indicate more difficulty.
Time Frame: Monthly up to one year
Population: Subsequent number of participants drops after baseline due to withdrawals or monthly follow-up not being completed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
units on a scale
  Baseline | 3.17 (3.005) | 3.46 (2.406)
  Month 1: number analyzed (Participants) | 68 | 64
  Month 1 | 2.79 (2.696) | 2.75 (2.397)
  Month 2: number analyzed (Participants) | 69 | 65
  Month 2 | 2.99 (2.841) | 3.05 (2.446)
  Month 3: number analyzed (Participants) | 67 | 65
  Month 3 | 2.96 (2.946) | 3.12 (2.362)
  Month 4: number analyzed (Participants) | 66 | 61
  Month 4 | 3.14 (2.762) | 3.34 (2.639)
  Month 5: number analyzed (Participants) | 64 | 64
  Month 5 | 3.45 (2.922) | 3.39 (2.741)
  Month 6: number analyzed (Participants) | 61 | 61
  Month 6 | 2.74 (2.613) | 2.95 (2.673)
  Month 7: number analyzed (Participants) | 62 | 58
  Month 7 | 2.95 (2.772) | 3.33 (2.691)
  Month 8: number analyzed (Participants) | 61 | 57
  Month 8 | 2.98 (2.723) | 3.07 (2.389)
  Month 9: number analyzed (Participants) | 59 | 58
  Month 9 | 2.98 (2.831) | 3.28 (2.821)
  Month 10: number analyzed (Participants) | 60 | 58
  Month 10 | 2.97 (2.414) | 3.14 (2.599)
  Month 11: number analyzed (Participants) | 59 | 59
  Month 11 | 2.90 (2.537) | 3.32 (2.381)
  Month 12: number analyzed (Participants) | 65 | 64
  Month 12 | 2.52 (2.599) | 2.58 (2.342)
Statistical Analysis 1: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Month 12 scores; Test type: Superiority; p = .900, t-test, 2 sided; Mean Difference (Net) = -0.055, 95% CI 2-sided [-0.917 to 0.807]

22. Secondary Outcome: Timed Loaded Standing Test
Description: A physical performance measure of combined trunk and arm endurance.
Time Frame: Baseline and one year
Population: Only participants from the University of Waterloo and the University of Toronto sites assessed.
Measure: Median (Standard Deviation); unit: Seconds
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 17 | 13
Seconds
  Baseline | 101.9 (39.8) | 107.5 (34.6)
  Month 12 | 120 (39.9) | 106 (37.6)
Statistical Analysis 1: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Baseline; Test type: Superiority; p = .712, t-test, 2 sided; Mean Difference (Final Values) = -5.2, 95% CI 2-sided [-33.6 to 23.2], Standard Error of Mean 13.9
Statistical Analysis 2: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Month 12; Test type: Superiority; p = .60, t-test, 1 sided; Mean Difference (Final Values) = 8.1, 95% CI 2-sided [-23.3 to 39.5], Standard Error of Mean 15.3

23. Secondary Outcome: Location of Vertebral Fractures
Description: Any vertebral fracture (Genant Grade 1 or higher) found on x-ray, divided into location groupings of T1-T3, T4-T8, T9-L1, and L2-L5.
Time Frame: Baseline and Month 12
Population: Withdrawals at 12 months - intervention group (n=5) and control group (n=6). The remainder (9 intervention, 8 control) did not have a second x-ray.
Measure: Number; unit: Fractures
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
Fractures
  Baseline T1-T3 | 3 | 1
  Baseline T4-T8 | 54 | 42
  Baseline T9-L1 | 74 | 88
  Baseline L2-L5 | 38 | 36
  Month 12 T1-T3: number analyzed (Participants) | 57 | 56
  Month 12 T1-T3 | 3 | 2
  Month 12 T4-T8: number analyzed (Participants) | 57 | 56
  Month 12 T4-T8 | 43 | 39
  Month 12 T9-L1: number analyzed (Participants) | 57 | 56
  Month 12 T9-L1 | 66 | 76
  Month 12 L2-L5: number analyzed (Participants) | 57 | 56
  Month 12 L2-L5 | 34 | 28

24. Secondary Outcome: Participant Weight
Time Frame: Baseline and Month 12
Population: Withdrawals at 12 months - intervention group (n=5) and control group (n=6). The remainder (7 intervention, 2 control) either did not attend the follow-up visit or did not have access to a scale at the visit.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
Number analyzed (Participants) | 71 | 70
kilograms
  Baseline | 65.1 (12.8) | 66.5 (15.4)
  Month 12: number analyzed (Participants) | 59 | 62
  Month 12 | 66.1 (13.3) | 66.6 (15.4)
Statistical Analysis 1: Comparison: Exercise and Behaviour Change Strategies vs General Health or Social Discussion; Comparison of change from baseline in weight; Test type: Superiority; p = 0.461, t-test, 2 sided; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.25 to 0.55] — Per-protocol analysis

ADVERSE EVENTS:
Arm/Group | Exercise and Behaviour Change Strategies | General Health or Social Discussion
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/70
Serious Adverse Events (participants affected / at risk) | 17/71 | 12/70
Other Adverse Events (participants affected / at risk) | 43/71 | 34/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise and Behaviour Change Strategies (N=71) | General Health or Social Discussion (N=70)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Idiopathic severe left foot pain (General disorders) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Adverse reaction to Forteo (Product Issues) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Dizziness (Cardiac disorders) | 1 (1) | 0 (0) — pulse was really slow and blood pressured dropped. Participant had a history of heart attack.
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Elevated blood pressure (Cardiac disorders) | 0 (0) | 1 (1) — palpitations and had very high blood pressure (220/110).
Severe vertigo (General disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Stomach infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vertebral pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extreme knee pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Shoulder dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise and Behaviour Change Strategies (N=71) | General Health or Social Discussion (N=70)
Irregular heart beat (Cardiac disorders) | 0 (0) | 2 (2)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Cataracts (Eye disorders) | 1 (2) | 0 (0)
Increased pain (General disorders) | 15 (20) | 5 (9)
Enlarged bile duct (Hepatobiliary disorders) | 0 (0) | 1 (1)
Rash (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
arthritis-related pains (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Bladder cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vaginal tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Obstructive sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Itchy scalp (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin basal cell carcinoma removed (Surgical and medical procedures) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Dizziness/loss of balance (General disorders) | 3 (3) | 0 (0)
Numbness/tingling in mouth (General disorders) | 2 (2) | 0 (0)
foot edema (General disorders) | 1 (1) | 0 (0)
corn infected on foot (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Infected finger (Infections and infestations) | 0 (0) | 1 (1)
Lyme Disease (Infections and infestations) | 1 (1) | 0 (0)
Meniere's Disease (Infections and infestations) | 1 (1) | 0 (0)
Pancreatitis (Infections and infestations) | 1 (2) | 0 (0)
Respiratory infection (Infections and infestations) | 4 (5) | 0 (0)
Shingles (Infections and infestations) | 3 (3) | 0 (0)
Sinus infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (4)
Fall/trip (Injury, poisoning and procedural complications) | 26 (29) | 12 (19)
Soft tissue injury (Injury, poisoning and procedural complications) | 4 (5) | 9 (11)
Domestic violence incident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Idiopathic breathing difficulties (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gallbladder Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder cyst surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Glass splinter removed from finger (Surgical and medical procedures) | 1 (2) | 0 (0)
Endoscopy (Surgical and medical procedures) | 0 (0) | 2 (2)
Facial growth removal (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No